CLINICAL TRIAL: NCT04859582
Title: A Phase 3, Randomized, Double-blind Clinical Study of Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy as First-line Treatment in Participants With HER2 Negative, Previously Untreated, Unresectable or Metastatic Gastric Orgastroesophageal Junction Adenocarcinoma (KEYNOTE-859)
Brief Title: Pembrolizumab (MK-3475) Plus Chemotherapy Versus Placebo Plus Chemotherapy in Participants Gastric or Gastroesophageal Junction (GEJ) Adenocarcinoma (MK-3475-859/KEYNOTE-859)-China Extension
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawn due to protocol amendment
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3475-859 China Extension; 2018-001757-27 (EudraCT Number); MK-3475-859 China Extension (Other: Merck); KEYNOTE-859 (Other: Merck); 194649 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2021-04-23; First posted 2021-04-26 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Stomach Neoplasms
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); programmed cell death ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pembrolizumab + FP or CAPOX (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5-fluorouracil (5FU) 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally twice a day (BID) on Days 1 to 14 Q3W. Participants who complete 35 administrations or achieve a complete response (CR) but progress after discontinuation can initiate a second course of pembrolizumab for up to 17 cycles (approximately 1 additional year).
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Capecitabine
- Placebo + FP or CAPOX (Active Comparator): Participants receive placebo for pembrolizumab IV on Day 1 Q3W for up to 35 cycles (approximately 2 years) + physicians' choice of either cisplatin 80 mg/m^2 IV on Day 1 Q3W and 5FU 800 mg/m^2/day via continuous IV infusion on Days 1 to 5 Q3W OR oxaliplatin 130 mg/m^2 IV on Day 1 Q3W + capecitabine 1000 mg/m^2 orally BID on Days 1 to 14 Q3W.
  Interventions: Drug: Cisplatin; Drug: 5-fluorouracil; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Placebo for Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered as an IV infusion on Day 1 Q3W
  Other Names: KEYTRUDA®; MK-3475
  Arms: Pembrolizumab + FP or CAPOX
Drug: Cisplatin — Administered as an IV infusion on Day 1 Q3W
  Other Names: PLATINOL®
Drug: 5-fluorouracil — Administered as a continuous IV infusion on Days 1-5 Q3W
  Other Names: ADRUCIL®; 5FU
Drug: Oxaliplatin — Administered as an IV infusion on Day 1 Q3W
  Other Names: ELOXATIN®
Drug: Capecitabine — Administered orally BID on Days 1 to 14 Q3W
  Other Names: XELODA®
Drug: Placebo for Pembrolizumab — Administered as an IV infusion on Day 1 Q3W
  Arms: Placebo + FP or CAPOX

SUMMARY:
The purpose of this study is to evaluate the efficacy of pembrolizumab (MK-3745) in combination with chemotherapy (Cisplatin combined with 5-Fluorouracil [FP regimen] or oxaliplatin combined with capecitabine [CAPOX regimen]) versus placebo in combination with chemotherapy (FP or CAPOX regimens) in the treatment of human epidermal growth factor receptor 2 (HER2) negative advanced gastric or GEJ adenocarcinoma in adult Chinese participants.

The primary hypotheses of this study are that pembrolizumab plus chemotherapy is superior to placebo plus chemotherapy in terms of overall survival (OS).

DETAILED DESCRIPTION:
The China extension study will include participants previously enrolled in China in the global study for MK-3475-859 (NCT03675737) plus those enrolled during the China extension enrollment period. A total of approximately 231 Chinese participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria

* Has histologically or cytologically confirmed diagnosis of locally advanced unresectable or metastatic gastric or gastroesophageal junction (GEJ) adenocarcinoma with known programmed cell death ligand 1 (PD-L1) expression status
* Has human epidermal growth factor receptor 2 (HER2) negative cancer
* Male participants must agree to use contraception during the intervention period and for at least 95 days after the last dose of chemotherapy, refrain from donating sperm and be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent or must agree to use contraception per study protocol unless confirmed to be azoospermic during this period
* Female participants who are not pregnant, not breastfeeding, and at least one of the following conditions applies: not a woman of childbearing potential (WOCBP) OR is a WOCBP who agrees to use contraception or be abstinent from heterosexual intercourse as their preferred and usual lifestyle during the treatment period and for at least 180 days after the last dose of chemotherapy or for at least 120 days after the last dose of pembrolizumab, whichever is last, and agrees not to donate eggs to others or freeze/store for her own use for the purpose of reproduction during this period
* Has measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator assessment
* Has provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated
* Has provided tumor tissue sample deemed adequate for PD-L1 biomarker analysis
* Has provided tumor tissue sample for microsatellite instability (MSI) biomarker analysis
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 3 days prior to the start of study intervention
* Has adequate organ function as demonstrated by laboratory testing within 10 days prior to the start of study treatment

Exclusion Criteria

* Has squamous cell or undifferentiated gastric cancer
* Has had major surgery, open biopsy, or significant traumatic injury within 28 days prior to randomization, anticipation of the need for major surgery during the course of study intervention, or has not recovered adequately from the toxicity and/or complications from previous surgery
* Has preexisting peripheral neuropathy >Grade 1
* Is a WOCBP who has a positive urine pregnancy test within 72 hours prior to randomization or treatment allocation
* Has had previous therapy for locally advanced, unresectable or metastatic gastric/GEJ cancer. Participants may have received prior neoadjuvant and/or adjuvant therapy as long as it was completed ≥6 months prior to randomization
* Has received prior therapy with an anti-PD-1, anti-PD-L1 or anti- PD-L2 agent or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), OX- 40, CD137)
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks prior to randomization or has not recovered from all AEs due to any previous therapies to ≤Grade 1 or baseline
* Has received prior radiotherapy within 2 weeks prior to study start or has not recovered from all previous radiation-related toxicities, required corticosteroids, and have not had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to noncentral nervous system (CNS) disease
* Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study treatment
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy
* Has known active CNS metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as Hepatitis C virus [HCV] ribonucleic acid [RNA] detected qualitatively) infection
* Has a known history of active tuberculosis
* Has hypokalemia (serum potassium less than the lower limit of normal)
* Has hypomagnesemia (serum magnesium less than the lower limit of normal)
* Has hypocalcemia (serum calcium less than the lower limit of normal)
* Has a history or current evidence of any condition (eg, known deficiency of the enzyme dihydropyrimidine dehydrogenase), therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of chemotherapy or through 120 days after the last dose of pembrolizumab, whichever is last
* Has had an allogenic tissue/solid organ transplant
* Has a known severe hypersensitivity (≥ Grade 3) to any of the study chemotherapy agents (including, but not limited to, infusional 5-fluorouracil or oral capecitabine) and/or to any of their excipients
* For participants taking cisplatin: has Grade ≥2 audiometric hearing loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-11-29 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 65 months
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 65 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR).
Objective Response Rate (ORR) | Up to approximately 65 months
  ORR was defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) | Up to approximately 65 months
  DOR is determined by disease assessment and is defined as the time from first response (CR or PR) to disease progression, or death from any cause, whichever occurs first.
Percentage of Participants Experiencing Adverse Events (AEs) | Up to approximately 65 months
  Percentage of participants experiencing an AE defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study therapy and irrespective of causality to study treatment.
Percentage of Participants Discontinuing Study Drug Due to AEs | Up to approximately 36 months
  Percentage of participants discontinuing study treatment due to an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (28):
- China (28):
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 2421), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 2425), Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital ( Site 2410), Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital ( Site 2414), Fuzhou, Fujian
  - 900 Hospital of the Joint ( Site 2418), Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University ( Site 2430), Xiamen, Fujian
  - Zhongshan Hospital Xiamen University ( Site 2447), Xiamen, Fujian
  - Guangdong General Hospital ( Site 2431), Guangzhou, Guangdong
  - Peking University Shenzhen Hospital ( Site 2442), Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 2401), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 2415), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 2434), Wuhan, Hubei
  - Xiangya Hospital Central-South University ( Site 2419), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 2439), Changsha, Hunan
  - Changzhou Cancer Hospital-Changzhou Fourth Peoples Hospital ( Site 2441), Changzhou, Jiangsu
  - The 81st Hospital of PLA ( Site 2413), Nanjing, Jiangsu
  - Jiangsu Cancer Hospital ( Site 2432), Nanjing, Jiangsu
  - Yancheng First People s Hospital ( Site 2426), Yancheng, Jiangsu
  - The First Affiliated Hospital of Nanchang University ( Site 2440), Nanchang, Jiangxi
  - The First Hospital of Jilin University ( Site 2416), Changchun, Jilin
  - The Affiliated Hospital of Qingdao University ( Site 2405), Qingdao, Shandong
  - Shanghai East Hospital ( Site 2403), Shanghai, Shanghai Municipality
  - Zhongshan Hospital affiliated to Fudan University ( Site 2407), Shanghai, Shanghai Municipality
  - 1st Affil hosp of Med College of Xi'an Jiaotong University ( Site 2428), XiAn, Shanxi
  - Cancer Hospital Affiliated to Xinjiang Medical University ( Site 2420), Ürümqi, Xinjiang
  - Zhejiang Provincial People's Hospital ( Site 2446), Hangzhou, Zhejiang
  - Sir Run Run Show Hospital ( Site 2427), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 2417), Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com